CLINICAL TRIAL: NCT01503151
Title: Cognitive Biases Modification Treatment for Social Anxiety
Acronym: CBMSP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Study Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: CBM_SP_2012
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Social Phobia
Keywords: attention bias modification treatment; interpretive bias modification; cognitive bias modification; attention training; social anxiety
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): repeated trials of a dot-probe task and repeated trials of an interpretation task, both not intended to change threat-related biases patterns.
  Interventions: Behavioral: Control Condition
- Attention Bias Modification (ABM) (Experimental): Attention training via repeated trials of a dot-probe task intended to direct attention away from threat stimuli.
  Interventions: Behavioral: Attention Bias Modification Treatment (ABMT)
- Interpretation Bias Modification (IBM) (Experimental): Interpretation training intended to facilitating a more benign interpretation bias
  Interventions: Behavioral: Interpretation Bias Modification (IBM)
- Attention and interpretation biases modification (Experimental): Attention and interpretation training intended to direct cognitive biases away from threat stimulus.
  Interventions: Behavioral: Attention and Interpretive biases modification (CBM)

INTERVENTIONS:
Behavioral: Attention Bias Modification Treatment (ABMT) — Attention training using a computerized spatial attention task (dot-probe) modified to alter threat-related attention patterns.
  Arms: Attention Bias Modification (ABM)
Behavioral: Interpretation Bias Modification (IBM) — Interpretive Bias Modification Treatment (IBMT) using a computerized task modified to facilitate a more benign interpretation bias.
  Arms: Interpretation Bias Modification (IBM)
Behavioral: Control Condition — Attention and interpretation training using a computerized tasks not intended to alter threat-related biases patterns.
  Arms: Placebo
Behavioral: Attention and Interpretive biases modification (CBM) — Attention and interpretation training via computerized tasks intended to direct attention away from threat stimuli and to facilitate a more benign interpretation bias.
  Arms: Attention and interpretation biases modification

SUMMARY:
Adults with Social Phobia will be randomly assigned to either an attention bias modification treatment, interpretation bias modification treatment, both, or a placebo control condition not designed to change cognitive bias patterns.

Outcome measures will be social anxiety symptoms and severity as measured by gold standard questionnaires as well as diagnosis of social phobia disorder and symptom counts derived from structured clinical interviews based on DSM-IV criteria.

The investigators expect to find significant reduction in social anxiety symptoms in the Treatment groups relative to the placebo control group. The investigators want to find out the relative efficacy of attention and interpretation oriented treatments and the combination of the two.

ELIGIBILITY:
Inclusion Criteria:

People suffering from social anxiety

Exclusion Criteria:

Pharmacological or Psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Social Anxiety Scale (LSAS) - diagnostic interview | Expected time frame of 6 weeks per participant. Participants will be assessed before and after the administration of the training/control protocols
  LSAS is a 24-items clinician-administered scale developed for the assessment of fear and avoidance associated with social. The LSAS assesses a wide range of both social interaction and performance/observation situations, which are rated for degree of fear/anxiety and frequency of avoidance.

SECONDARY OUTCOMES:
The Mini International Neuropsychiatric Interview (MINI). | expected time frame of 6 weeks per participant. Participants will be assessed before and after the administration of the training/control protocols
  The Mini International Neuropsychiatric Interview (MINI) is a short diagnostic structured interview (DSI) developed to explore 17 disorders according to Diagnostic and Statistical Manual diagnostic criteria (DSM)

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel